CLINICAL TRIAL: NCT06647498
Title: A Phase II/III Multicenter Randomized, Double-Blind, Placebo-Controlled, Two-Stage Adaptive Design, Platform Trial of Investigational Treatments for Primary Prevention of Disease Progression in Dominantly Inherited Alzheimer's Disease
Brief Title: A Study of a Potential Disease Modifying Treatment in Individuals at Risk for or With a Type of Early Onset AD Caused by a Genetic Mutation
Acronym: DIAN-TU-002
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Alzheimer's Association (Other); Eli Lilly and Company (Industry); National Institute on Aging (NIA) (NIH); GHR Foundation (Unknown); Private Donors (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAN-TU-002 (REM); 5U01AG059798 (NIH)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alzheimers Disease; Dementia; Alzheimers Disease, Familial
Keywords: Alzheimer's; Alzheimer's Disease; Dementia; Mutation; Genetic Mutation; Dominantly Inherited Alzheimer's Disease; Dominantly Inherited Alzheimer Network; Autosomal Dominant Alzheimer's Disease; Early Onset Alzheimer's Disease; DIAN; DIAN-TU; DIAN TU; DIAD
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Stage 1: Interventional/matching placebo; Stage 2: Open Label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stage 1: Remternetug (Experimental): Active Remternetug- blinded
  Interventions: Drug: Remternetug
- Stage 1: Matching placebo (Remternetug) (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching Placebo (Remternetug)
- Stage 2: Remternetug Open Label (Active Comparator): Open label will start after last dose of Stage 1

INTERVENTIONS:
Drug: Remternetug — Administered subcutaneously every 12 weeks
  Other Names: LY3372993
  Arms: Stage 1: Remternetug
Drug: Matching Placebo (Remternetug) — Administered as subcutaneous injection of placebo every 12 weeks
  Arms: Stage 1: Matching placebo (Remternetug)

SUMMARY:
The purpose of this research study is to test the study drug, referred to as remternetug, to determine its effectiveness for the study treatment of asymptomatic (at risk) Alzheimer disease in individuals with AD-causing mutations. This study will also investigate the effects of remternetug on biomarkers (measures of the disease including brain scans, blood and spinal fluid tests), examine safety data to identify any potential benefits or risks, and examine how well participants can tolerate remternetug.

Stage 1 will determine if treatment with the study drug prevents or reverses amyloid beta (Aβ) accumulation compared with placebo in participants with dominantly inherited Alzheimer's disease (DIAD).

Stage 2 will evaluate the effect of early anti-amyloid treatment on downstream biomarkers of AD in treated participants compared to external control groups.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is an age-related neurodegenerative disorder characterized by progressive decline in cognitive function and the ability to perform activities of daily living. The amyloid hypothesis of AD postulates that the accumulation of amyloid beta (Aβ) is an early and necessary event in the pathogenesis of AD. This hypothesis suggests that interventions that slow the accumulation of Aβ plaque in the brain or increase clearance of Aβ may be able to slow the progression of the AD clinical syndrome. AD occurs on a continuum from asymptomatic (preclinical) to mild cognitive impairment (MCI), and then to dementia in mild, moderate, and severe stages. Evidence from both genetic at-risk and age at-risk cohorts, such as in dominantly inherited AD (DIAD) suggests that the pathophysiological process of AD begins well more than a decade before the clinical stage now recognized as AD dementia, and that neurodegeneration is already apparent on MRI by the stage of mild cognitive impairment. Recent clinical trial data suggest that treating AD during the earlier stages could have the greatest potential benefit on the disease by slowing progression

The ability to identify individuals destined to develop Alzheimer's disease (AD) with a high degree of confidence provides a unique opportunity to assess the efficacy of therapies at asymptomatic and very early stages of dementia. Families with known disease-causing mutations are extremely rare and are geographically dispersed throughout the world.

Participants in this study will not yet have developed any clinical symptoms of AD; they will be "asymptomatic" carriers of mutations that cause DIAD and would be expected to perform normally on standard cognitive and functional testing. Further, most mutation carriers will have levels of AD-associated amyloid beta (Aβ) and non-Aβ biomarkers that are the same as non-carriers.

Amyloid beta is a protein that accumulates in the brain of people with AD. Although we do not understand exactly what causes AD, the abnormal accumulation of amyloid beta protein in the brain is thought to play an important role in the symptoms of AD. Recent research studies indicate that amyloid beta may start building up in the brain 15 years or more before the onset of memory loss.

Imaging and fluid biomarkers will be used to demonstrate that the treatment compounds have engaged their therapeutic targets. A set of cognitive measures designed to assess the very earliest and most subtle cognitive changes will be collected. The overall objectives of this study are to evaluate the biomarker effect, safety, and tolerability of investigational study drugs in participants who are known to have an AD-causing mutation.

The primary objective of Stage 1 is to determine if treatment with the study drug prevents or slows the rate of Aβ pathological disease accumulation demonstrated by Aβ PiB positron emission tomography (PET) imaging.

The primary objective of Stage 2 is to evaluate the effect of early anti-amyloid treatment on disease progression by assessing downstream non-Aβ biomarkers of AD (e.g., CSF total tau, NfL, MRI volume) compared to a control group from the DIAN Obs natural history study and the DIAN-TU-001 placebo-treated participants.

Remternetug is a monoclonal antibody. The mechanism of action of remternetug is to target and remove aggregated amyloid plaque, a key pathological hallmark of AD, via microglial-mediated clearance. Remternetug has demonstrated the ability to reduce brain amyloid plaque.

The remternetug arm is part of Master Protocol DIAN-TU-002 (NCT05552157)

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, signed, and dated by the participant and study partner, or by the participant's legally authorized representative if applicable, according to local regulations for the ICF and, if applicable, country specific ICFs.
2. Participant is at least 18 years old.
3. People of childbearing potential

   1. Must have a negative serum pregnancy test at screening (V1)
   2. Must agree not to try to become pregnant during the study until 5 half-lives after the last dose of any study drug.
   3. Must agree not to breastfeed from the time of signed ICF until 5 half-lives after the last dose of any study drug.
   4. If partner is not sterilized, must agree to use highly effective contraceptive measures from screening (V1) until 5 half lives after last dose of any study drug
4. Mutation Status:

   1. Participant is a carrier of a mutation in an APP, PSEN1, or PSEN2 gene that is associated with DIAD or does not know their mutation status and there is a mutation in their family pedigree that puts them at a direct risk of inheriting the known mutation;
   2. Participant is -25 to -11 years from predicted age of cognitive symptom onset based on their mutation type or family pedigree Note: If the at-risk parent is deemed a non-carrier through confirmed genetic testing at any time during the study, the participant will be withdrawn.
5. Cognitive status of participant is normal (CDR-SB 0).
6. Fluency in DIAN-TU trial approved language and evidence of adequate premorbid intellectual functioning. Participants must be fluent in languages for which cognitive and clinical measures have been translated and validated for use in the DIAN-TU. Fluency is generally defined as daily or frequent functional use of a language generally from birth or a young age. In cultures where multiple languages are spoken or for participants who are multilingual, determination as to whether a participant's level of fluency in languages for which clinical and cognitive measures are available meets qualification for the study should be made by the site PI.
7. Participant has adequate visual and auditory abilities to perform all aspects of the cognitive and clinical assessments.
8. Participant is receiving stable doses of medication(s) for the treatment of non-excluded medical condition(s) for at least 30 days prior to baseline visit (V2) except for medications taken for episodic conditions (e.g., migraine abortive therapy, antibiotics, and other medications for upper respiratory and gastrointestinal ailments).
9. Participant has a study partner who in the PI's judgment can provide accurate information as to the participant's cognitive and functional abilities, who agrees to provide information at the study visits that require study partner input for scale completion, and who signs the necessary ICF, if applicable.
10. The participant agrees not to donate blood or blood products for transfusion from the time of Screening (V1) for a study drug arm, for the duration of the study, and for 5 half lives after the final dose of study drug.
11. In the opinion of the PI, the participant will be compliant and have a high probability of completing the study.
12. The participant is able and willing to complete all study-related testing, evaluations, and procedures.

Exclusion Criteria:

1. Significant neurologic disease (other than AD) or psychiatric disease that may currently or during the study affect cognition or the participant's ability to complete the study. This would include disorders such as: recent or severe head trauma causing cognitive change, seizure disorder, neurodegenerative disease other than DIAD, hydrocephalus, cerebral/spinal hematoma, inflammatory disease, CNS infection (e.g., encephalitis or meningitis), neoplasm, toxic exposure, metabolic disorder (including hypoxic or hypoglycemic episodes) or endocrine disorder; psychiatric disorders such as schizophrenia, schizoaffective disorder, bipolar disorder or major depression, or any other psychiatric condition/disorder which could significantly interfere with the participant's cooperative participation (e.g., prominent anxiety, agitation or behavioral problems). Disorders that are controlled medically or remote history of these disorders (e.g., history of febrile seizures in childhood) that are not likely to interfere with cognitive function and compliance with study procedures are not exclusionary.
2. At high risk for suicide, e.g., significant suicidal ideation or attempt within last 12 months, current major depression (as defined in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-V]), or increased suicide risk based on screening Columbia Suicide Severity Rating Scale (C-SSRS). Current stable mild depression or current use of antidepressant medications are not exclusionary.
3. History of clinically evident stroke or history of clinically important carotid or vertebrobasilar stenosis, plaque, or other prominent risk factor for stroke or cerebral hemorrhage (including atrial fibrillation and anticoagulation, documented transient ischemic attack [TIA] in the last 12 months) that may be interfering with cognition or is likely to impact with the participant's ability to complete the study. Low dose aspirin (≤ 325 mg daily) is not exclusionary.
4. Alcohol or substance use sufficient to meet DSM-V criteria currently or within the past year.
5. History of or Baseline (V2) visit brain MRI scan indicative of any other significant abnormality, definite microhemorrhages, evidence of a cerebral contusion, encephalomalacia, or aneurysms. Minor or clinically insignificant imaging findings are not exclusionary.
6. Presence of certain implanted medical devices, such as some pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body which would preclude MRI scan.
7. Cardiovascular complications such as uncontrolled hypertension, history of myocardial infarcts, heart failure, atrial fibrillation, long QT interval on ECG likely to interfere with participation in or analysis of the trial in the opinion of the investigator
8. Hepatic or renal abnormalities that in the opinion of the investigator would interfere with participation in or analysis of the trial.
9. History of Human Immunodeficiency Virus (HIV) infection, history of Hepatitis B infection within the past year, history of Hepatitis C infection which has not been adequately treated, history of spirochete infection (e.g., syphilis, Lyme) of the CNS or history of other infection with high risk for interfering with participation or interpretation of the study in the opinion of the investigator.
10. History of clinically significant multiple or severe drug allergies, significant atopy, or severe post-treatment hypersensitivity reactions (including but not limited to erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, and/or exfoliative dermatitis) or sensitivity to study-drug specific PET imaging agents with a high risk for interfering with participation or interpretation of the study in the opinion of the investigator.
11. Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within 90 days prior to Baseline (V2) visit (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years.
12. Current clinically significant abnormalities of thyroid function, or clinically significant deficiency in vitamin B12. Vitamin B12 less than the lower limits of normal with normal methylmalonic acid (MMA)/homocysteine is not deemed clinically significant, therefore not exclusionary.
13. Unstable or poorly controlled diabetes which the investigator believes may interfere with participation in or analysis of the study protocol. Participants may be rescreened after 3 months to allow optimization of diabetic control
14. Morbid obesity with significant comorbidities or that would preclude MRI imaging.
15. Current use of anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, or apixaban). Daily use of low dose (< 325 mg) aspirin is not exclusionary.
16. Have been exposed to a monoclonal antibody targeting Aβ peptide within the past 6 months or 5 half-lives from screening, whichever is longer.
17. Received any other investigational pharmacological treatment within 3 months of Screening or 5 half-lives, whichever is longer.

    Note: Use of approved treatments for AD and other medications may be permitted in this study.
18. Lack of sufficient venous access.
19. Clinically relevant abnormalities in hematology, coagulation, or clinical chemistry.
20. History of cancer that the investigator believes has high risk of recurrence and impacting study participation or analysis.
21. Any other medical condition that could be expected to progress, recur, or change to such an extent that it could bias the assessment of the clinical or mental status of the participant to a significant degree or put the participant at special risk.
22. Currently, or within the last month prior to screening, participated in a clinical study, including a nonpharmacological study, without prior approval.
23. Participants with the "Dutch" APP E693Q mutation.
24. Unable to complete baseline visit (V2) procedures with appropriate cognitive and clinical scores for eligibility
25. A centrally read MRI demonstrating presence of ARIA-E, > 4 cerebral microhemorrhages, any superficial siderosis, any macrohemorrhage, or severe white matter disease at screening.
26. Exposure to lecanemab, donanemab, or other investigational amyloid lowering agents within the past 6 months or five half-lives from screening, whichever is longer.

    Note: Use of approved treatments for AD and other medications may be permitted.
27. Investigator site personnel directly affiliated with this trial and/or their immediate families, defined as a spouse, parent, child, or sibling, whether biological or legally adopted
28. Lilly employees or employees of a third-party organization (TPO) involved in this study that requires exclusion of their employees or have study partners who are Lilly employees or are employees of TPOs involved in this study that require exclusion of their employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2034-03 (Estimated); Study Completion 2034-08 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Change in amyloid load as measured by centiloid (CL) [11C]PiB-PET as biomarker endpoint for DIAN-TU-002 remternetug arm | Baseline and Week 192
  CL calculated using [11C] PiB PET non-partial volume corrected (regional spread function) standardized uptake value ratio cortical composite (PiB PET SUVR) is the primary outcome and change from baseline at 2 years is the primary endpoint.

SECONDARY OUTCOMES:
Stage 2: Odds ratio between the drug-treated and control groups of being in the lower biomarker disease progression stage based on two-stage modeling of 6 biomarkers. | Weeks 0, 48, 96, 144, and 192
  The key secondary efficacy endpoint for Stage 2 is the odds ratio between the treated group and the external control group (DIAN Obs and DIAN-TU-001 placebo) of being in the lower biomarker disease progression stage based on two-stage modeling of 6 biomarkers (CSF tau phosphorylated tau at residue 153 (pTau153)/Tau153 ratio, CSF pTau205/Tau205 ratio, CSF microtubule binding region of tau 243 amino acids long (MTBR-tau243), MRI hippocampal volume, CSF neurofilament light chain (NfL), and MRI precuneus thickness).
Stage 1: The proportion of participants who are amyloid positive (CL level ≥ 16.3) at the end of Stage 1 | Baseline and Week 104
  For participants in the active treatment group, the amyloid positivity status is defined using the last available PiB-PET CL value during Stage 1: amyloid positive if CL>=16.3 and amyloid negative if CL<16.3. For participants in the placebo group, the amyloid positivity status: (i) is either defined using the last available PiB-PET CL value during Stage 1 (amyloid positive if CL>=16.3 and amyloid negative if CL<16.3)
Stage 1: Change in CSF pTau217/Tau217 ratio | Baseline and Week 104
Stage 1: Change in CSF pTau231/Tau231 ratio | Baseline and week 104
Stage 1: Change in CSF 3-repeat isoform of MTBR (MTBR-3R) | Baseline and week 104
Stage 2: Change in CSF pTau217/Tau217 ratio CSF pTau231/Tau231 ratio, and CSF MTBR-3R | Weeks 0, 48, 96, 144, and 192
Stage 2: Change in Cognitive Composite Score | Weeks 0, 48, 96, 144, and 192
  A cognitive composite derived as an average of these four tests: Memory Complaint Questionnaire (MAC-Q), Category Fluency (Animals), Buschke and Grober Free and Cued Selective Reminding Test - Immediate Recall (FCSRT-IR), Wechsler Adult Intelligence Scale - Revised (WAIS-R) Digit Symbol Substitution Test, and Mini-Mental State Examination (MMSE). Each of the four tests will be converted to a z-score using the mean (SD) of the baseline score in Stage 1 of both the treatment arm and the placebo arm, and then equally weighted to obtain the composite.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M McDade, DO, Study Director — Washington University School of Medicine
Locations (35):
- United States (12):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Kerwin Research and Memory Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- Instituto de Investigaciones Neurologicas Raul Carrea, FLENI, Ciudad Autonoma de Buenos Aire, Argentina
- Australia (2):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Mental Health Research Institute, Melbourne, Victoria
- Canada (4):
  - UBC Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill Center for Studies in Aging, Verdun, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Grupo de Neurociencias Sede de la Universidad de Antioquia, Medellín, Colombia
- France (5):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
- Germany (2):
  - Universitaetsklinikum Tubingen, Tübingen, Baden-Wurttemberg
  - LMU-Campus Grosshadern, Munich, Bavaria
- Italy (2):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
- Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez, Mexico City, Mexico City, Mexico
- Brain Research Center, Amsterdam, Netherlands
- New Zealand Brain Research Institute, Christchurch, New Zealand
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico, Puerto Rico
- Hospital Clínic I Provincial de Barcelona, Barcelona, Barcelona, Spain
- The National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to DIAN-TU trial data will follow the DIAN-TU data access policy, which complies with the guidelines established by the Collaboration for Alzheimer's Prevention [CAP REF].
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] McDade E, Bateman RJ. Tau Positron Emission Tomography in Autosomal Dominant Alzheimer Disease: Small Windows, Big Picture. JAMA Neurol. 2018 May 1;75(5):536-538. doi: 10.1001/jamaneurol.2017.4026. No abstract available. PMID 29435570
- [Background] Fagan AM, Xiong C, Jasielec MS, Bateman RJ, Goate AM, Benzinger TL, Ghetti B, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Salloway S, Schofield PR, Sperling RA, Marcus D, Cairns NJ, Buckles VD, Ladenson JH, Morris JC, Holtzman DM; Dominantly Inherited Alzheimer Network. Longitudinal change in CSF biomarkers in autosomal-dominant Alzheimer's disease. Sci Transl Med. 2014 Mar 5;6(226):226ra30. doi: 10.1126/scitranslmed.3007901. PMID 24598588
- [Background] Fagan AM, Roe CM, Xiong C, Mintun MA, Morris JC, Holtzman DM. Cerebrospinal fluid tau/beta-amyloid(42) ratio as a prediction of cognitive decline in nondemented older adults. Arch Neurol. 2007 Mar;64(3):343-9. doi: 10.1001/archneur.64.3.noc60123. Epub 2007 Jan 8. PMID 17210801
- [Background] Demattos RB, Lu J, Tang Y, Racke MM, Delong CA, Tzaferis JA, Hole JT, Forster BM, McDonnell PC, Liu F, Kinley RD, Jordan WH, Hutton ML. A plaque-specific antibody clears existing beta-amyloid plaques in Alzheimer's disease mice. Neuron. 2012 Dec 6;76(5):908-20. doi: 10.1016/j.neuron.2012.10.029. PMID 23217740
- [Background] Young AL, Oxtoby NP, Daga P, Cash DM, Fox NC, Ourselin S, Schott JM, Alexander DC; Alzheimer's Disease Neuroimaging Initiative. A data-driven model of biomarker changes in sporadic Alzheimer's disease. Brain. 2014 Sep;137(Pt 9):2564-77. doi: 10.1093/brain/awu176. Epub 2014 Jul 9. PMID 25012224
- [Background] Sims JR, Zimmer JA, Evans CD, Lu M, Ardayfio P, Sparks J, Wessels AM, Shcherbinin S, Wang H, Monkul Nery ES, Collins EC, Solomon P, Salloway S, Apostolova LG, Hansson O, Ritchie C, Brooks DA, Mintun M, Skovronsky DM; TRAILBLAZER-ALZ 2 Investigators. Donanemab in Early Symptomatic Alzheimer Disease: The TRAILBLAZER-ALZ 2 Randomized Clinical Trial. JAMA. 2023 Aug 8;330(6):512-527. doi: 10.1001/jama.2023.13239. PMID 37459141
- [Background] Oxtoby NP, Young AL, Cash DM, Benzinger TLS, Fagan AM, Morris JC, Bateman RJ, Fox NC, Schott JM, Alexander DC. Data-driven models of dominantly-inherited Alzheimer's disease progression. Brain. 2018 May 1;141(5):1529-1544. doi: 10.1093/brain/awy050. PMID 29579160
- [Background] Navitsky M, Joshi AD, Kennedy I, Klunk WE, Rowe CC, Wong DF, Pontecorvo MJ, Mintun MA, Devous MD Sr. Standardization of amyloid quantitation with florbetapir standardized uptake value ratios to the Centiloid scale. Alzheimers Dement. 2018 Dec;14(12):1565-1571. doi: 10.1016/j.jalz.2018.06.1353. Epub 2018 Jul 11. PMID 30006100
- [Background] Hardy J, Selkoe DJ. The amyloid hypothesis of Alzheimer's disease: progress and problems on the road to therapeutics. Science. 2002 Jul 19;297(5580):353-6. doi: 10.1126/science.1072994. PMID 12130773
- [Background] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Background] Rabinovici GD, Furst AJ, Alkalay A, Racine CA, O'Neil JP, Janabi M, Baker SL, Agarwal N, Bonasera SJ, Mormino EC, Weiner MW, Gorno-Tempini ML, Rosen HJ, Miller BL, Jagust WJ. Increased metabolic vulnerability in early-onset Alzheimer's disease is not related to amyloid burden. Brain. 2010 Feb;133(Pt 2):512-28. doi: 10.1093/brain/awp326. Epub 2010 Jan 15. PMID 20080878
- [Background] Price JL, McKeel DW Jr, Buckles VD, Roe CM, Xiong C, Grundman M, Hansen LA, Petersen RC, Parisi JE, Dickson DW, Smith CD, Davis DG, Schmitt FA, Markesbery WR, Kaye J, Kurlan R, Hulette C, Kurland BF, Higdon R, Kukull W, Morris JC. Neuropathology of nondemented aging: presumptive evidence for preclinical Alzheimer disease. Neurobiol Aging. 2009 Jul;30(7):1026-36. doi: 10.1016/j.neurobiolaging.2009.04.002. Epub 2009 Apr 18. PMID 19376612
- [Background] Price JL, Morris JC. Tangles and plaques in nondemented aging and "preclinical" Alzheimer's disease. Ann Neurol. 1999 Mar;45(3):358-68. doi: 10.1002/1531-8249(199903)45:33.0.co;2-x. PMID 10072051
- [Background] Mills SM, Mallmann J, Santacruz AM, Fuqua A, Carril M, Aisen PS, Althage MC, Belyew S, Benzinger TL, Brooks WS, Buckles VD, Cairns NJ, Clifford D, Danek A, Fagan AM, Farlow M, Fox N, Ghetti B, Goate AM, Heinrichs D, Hornbeck R, Jack C, Jucker M, Klunk WE, Marcus DS, Martins RN, Masters CM, Mayeux R, McDade E, Morris JC, Oliver A, Ringman JM, Rossor MN, Salloway S, Schofield PR, Snider J, Snyder P, Sperling RA, Stewart C, Thomas RG, Xiong C, Bateman RJ. Preclinical trials in autosomal dominant AD: implementation of the DIAN-TU trial. Rev Neurol (Paris). 2013 Oct;169(10):737-43. doi: 10.1016/j.neurol.2013.07.017. Epub 2013 Sep 6. PMID 24016464
- [Background] McDade E, Wang G, Gordon BA, Hassenstab J, Benzinger TLS, Buckles V, Fagan AM, Holtzman DM, Cairns NJ, Goate AM, Marcus DS, Morris JC, Paumier K, Xiong C, Allegri R, Berman SB, Klunk W, Noble J, Ringman J, Ghetti B, Farlow M, Sperling RA, Chhatwal J, Salloway S, Graff-Radford NR, Schofield PR, Masters C, Rossor MN, Fox NC, Levin J, Jucker M, Bateman RJ; Dominantly Inherited Alzheimer Network. Longitudinal cognitive and biomarker changes in dominantly inherited Alzheimer disease. Neurology. 2018 Oct 2;91(14):e1295-e1306. doi: 10.1212/WNL.0000000000006277. Epub 2018 Sep 14. PMID 30217935
- [Background] Ryman DC, Acosta-Baena N, Aisen PS, Bird T, Danek A, Fox NC, Goate A, Frommelt P, Ghetti B, Langbaum JB, Lopera F, Martins R, Masters CL, Mayeux RP, McDade E, Moreno S, Reiman EM, Ringman JM, Salloway S, Schofield PR, Sperling R, Tariot PN, Xiong C, Morris JC, Bateman RJ; Dominantly Inherited Alzheimer Network. Symptom onset in autosomal dominant Alzheimer disease: a systematic review and meta-analysis. Neurology. 2014 Jul 15;83(3):253-60. doi: 10.1212/WNL.0000000000000596. Epub 2014 Jun 13. PMID 24928124
- See also: Expanded registry — http://www.dianexr.org/